CLINICAL TRIAL: NCT01029665
Title: Early Childhood Follow-up of Congenital Diaphragmatic Hernia Survivors
Acronym: CDH
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00006486; 392-1577 (Other Grant/Funding Number: Discovery Labs)
Record Dates: First submitted 2009-11-19; First posted 2009-12-10 (Estimated); Last update posted 2024-04-12 (Actual); Status verified 2013-03

CONDITIONS: Hernia, Diaphragmatic
Keywords: Hernia, Diaphragmatic; Asthma; Feeding and Eating Disorders of Childhood; Growth & Development
MeSH Terms: conditions — Hernia, Diaphragmatic; Asthma; Feeding and Eating Disorders of Childhood

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CDH survivors: School age (ages 4-6) Congenital Diaphragmatic Hernia survivors treated at Duke University Medical Center.

SUMMARY:
The primary objective of this study is to determine the medical and neurodevelopmental outcomes of congenital diaphragmatic hernia (CDH) survivors at school-age (4-6 years) follow-up. It is generally assumed that older CDH survivors have normal daily function and are able to live normal lives, but this has not been adequately studied.

DETAILED DESCRIPTION:
Congenital diaphragmatic hernia (CDH) is a relatively rare malformation, seen in approximately 1 in 3000-5000 live births. The overall survival for infants born with CDH ranges from 50-70% despite continuing advances in prenatal diagnosis and post-natal medical and surgical care. Infants with CDH remain one of the most complex groups of patients to care for - both in the intensive care nursery and after hospital discharge.

Several studies have shown that CDH survivors have predictable pulmonary, gastrointestinal, cardiac, and neurologic morbidities. In particular, CDH survivors are at an increased risk for growth and nutrition difficulties, including feeding problems, symptomatic gastroesophageal reflux, and failure to thrive. They are also more likely to suffer from chronic lung disease, bronchial hyperreactivity, and pulmonary hypertension. In addition, a significant number of CDH survivors show evidence of neurocognitive delay, hearing impairment, and behavioral disorders in follow-up studies.

Most outcome studies of CDH survivors have focused on the 18-36 month follow-up period. However, there is a paucity of literature on longer-term, school-age outcomes of these children. In order that we might better understand the impact of our current CDH management protocols, it is imperative to determine whether the cognitive delays and other morbidities noted in these patients at an early age are of a transient nature, or persist throughout childhood. It is also crucial to develop a predictive model to understand which patients with CDH will undoubtedly develop long-term neurodevelopmental impairment. Collecting and sharing knowledge with the broader community of Neonatal Intensive Care providers who manage infants with CDH will ultimately help guide therapeutic strategies in the intensive care nursery so that parents can make informed decisions about aggressiveness of care and we may optimize the outcomes of this unique patient population.

ELIGIBILITY:
Inclusion Criteria:

* Survivors of CDH who are at least 4 years old at the time of the study will be eligible for inclusion in the follow-up portion of the study.

Exclusion Criteria:

* Spanish-speaking only children and families.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All infants with Congenital Diaphragmatic Hernia (CDH) born between 2001 and 2005 who were managed at Duke University Medical Center will be eligible for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2008-09; Primary Completion 2009-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Persistent medical morbidities and/or neurodevelopmental impairment at school age (ages 4-6). | Visit 1

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer R Benjamin, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States